CLINICAL TRIAL: NCT03241836
Title: Role of Trans-perineal Ultrasonography on Basis of Dynamic Pelvic Magnetic Resonance Imaging in Diagnosis of Female Pelvic Floor Dysfunction
Brief Title: Trans-perineal Ultrasound & Dynamic Pelvic Magnetic Resonance Imaging in Assessment of Pelvic Floor Dysfunction.
Status: Withdrawn | Type: Observational
Why Stopped: 3Dtransvaginal probe is not available at this time
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, AShassan, principle investigator, Assiut University
Other Study IDs: TPUS& MRI female pelvic floor
Record Dates: First submitted 2017-08-01; First posted 2017-08-08 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Floor, Obstetric

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: trans-perineal ultrasonography — accuracy of trans perineal ultrasonography in identification of female pelvic floor dysfunction
  Other Names: dynamic pelvic MRI

SUMMARY:
Pelvic floor failure is a common disorder that can seriously jeopardize woman's quality of life by causing urinary, fecal incontinence, difficult defecation and pelvic pain. Multiple congenital and acquired risk factors are associated with pelvic floor failure including altered collagen metabolism, female sex, vaginal delivery, menopause, and advanced age. A complex variety of fascial and muscular lesions that range from stretching, insertion detachment, denervation atrophy, and combinations of pelvic floor relaxation to pelvic organ prolapse may manifest in a single patient.

The prevalence of pelvic floor dysfunction increases with age. It is approximately 9.7% in child bearing period (20-39 yrs), while it reaches up to 49.7% by 80 yrs and older.

Thorough preoperative assessment of pelvic floor failure is necessary to reduce the rate of relapse, which is reported to be as high as 30%.

MR imaging is a powerful tool that enables radiologists to comprehensively evaluate pelvic anatomic and functional abnormalities, thus helping surgeons provide appropriate treatment and avoid repeat operations.

Real time 2D trans-perineal ultrasound is emerging as an exciting new technique for pelvic floor assessment. It has advantage of providing a global view of the entire pelvic floor, from the symphysis to the ano-rectum, and includes the lower aspects of the levator ani muscle, in addition to its lower costs and greater accessibility; also sonographic imaging is more useful in the clinical environment, and generally better tolerated than MRI.

DETAILED DESCRIPTION:
135 female patients in child bearing period (20-39 yrs) will undergo trans-perineal US and dynamic pelvic MRI; 40 days after vaginal delivery or cesarean section for asymptomatic and symptomatic cases.

Revision after six months for cases with sonongraphic or MRI findings. after obtaining an informed written consent and approval of the ethical committee of faculty of medicine of Assiut University.

* Inclusion criteria: asmptomatic and symptomatic female Patients in child bearing period 40 days after vaginal delivery and cesarean section.
* Exclusion criteria: patients with previous pelvic floor surgery.

Patient preparation

For trans-perineal US:

- Patient is positioned in dorsal lithotomy position, with the hips flexed and slightly abducted and after bladder and bowel emptying. The pelvic tilt can be improved by asking the patient to place their heels as close as possible to the but¬tocks and move hips towards the heels.

For MRI:

- Patient is positioned in supine position and using pelvic coil after bladder and bowel emptying.

Method:

1. trans-perineal US: B mode capable 2D ultrasound system with cine loop function, 3.5-6.0 MHz curved array transducer. A mid-sagittal and axial views is obtained by placing a transducer on the perineum (Parting of the labia can improve image quality).
2. Dynamic MRI:

Magnetic resonance (MR) imaging of the pelvic floor is a two-step process that includes:

Analysis of anatomic damage on axial, coronal and sagittal fast spin-echo (FSE) T2-weighted images.

Functional evaluation using sagittal dynamic single-shot T2-weighted sequences during straining and defecation.

ELIGIBILITY:
* Inclusion criteria: asmptomatic and symptomatic female Patients in child bearing period 40 days after vaginal delivery and cesarean section.
* Exclusion criteria: patients with previous pelvic floor surgery.

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: female patients in child bearing period (20-39 yrs old) with or without symptoms of pelvic floor failure
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
accuracy of trans-perineal ultrasonography in assessment of pelvic floor dysfunction | four years

CONTACTS AND LOCATIONS:
Overall Officials: alzahraa sayed hassan, a.lecturer, Principal Investigator — Assiut University